CLINICAL TRIAL: NCT06170294
Title: A Single-arm, Open-label, Dose Exploratory Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of Autologous Humanized MAGE-A4-directed T Cell Receptor Engineered T Cell (JWTCR001) in Patients With Advanced Solid Tumors
Brief Title: MAGE-A4-directed TCR-T in the Treatment Amongst Subjects With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: Shanghai Ming Ju Biotechnology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Shen Lin, Professor, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JWTCR001001
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TCR-MAGE-A4 T-Cells (Experimental): The subjects enrolled will be sequentially assigned to the corresponding dose level.
  Interventions: Drug: TCR-MAGE-A4 T-Cells

INTERVENTIONS:
Drug: TCR-MAGE-A4 T-Cells — * Preconditioning with fludarabine, cyclophosphamide, based chemotherapy regimen at sub-clinical doses
  * MAGE-A4-directed T cell receptor-engineered T Cells
  Other Names: MAGE-A4-directed T cell receptor-engineered T Cells

SUMMARY:
A single-arm, open-label, dose exploratory study to evaluate the safety, efficacy, and pharmacokinetics of autologous humanized anti-MAGE-A4 T cell receptor-engineered T cell (TCR-T) in advanced solid tumors.

DETAILED DESCRIPTION:
This study is a single-arm, open-label, dose escalation/dose regimen finding study to assess the safety and pharmacokinetics of T-cell receptor-engineered T cell (TCR-T) targeting melanoma-associated antigen-4 (MAGE-A4) and to obtain the preliminary efficacy results in subjects who have been diagnosed with advanced solid tumors with positive MAGE-A4 expression and refractory to prior standard systemic treatments.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 year-old, male or female
2. Voluntarily willing to participate in the study and sign the written informed consent form
3. Life expectation ≥12 weeks
4. European Cooperative Oncology Group (ECOG) ≤1 at screening, 24 hours prior to apheresis (APH), lymphodepletion (LD), and infusion
5. Histologically-confirmed recurrent/metastatic advanced solid tumors
6. Radiologically-confirmed progression disease after at least one prior line of systematic treatment and no available standard of care at screening, judged by investigators
7. Fresh or formalin-fixed paraffin-embedded (FFPE) samples, immunohistochemistry (IHC)-stained MAGE-A4 positive
8. Human leukocyte antigen (HLA)-A*02 allele matched
9. Per response evaluation criteria in solid tumors (RECIST) version 1.1, at least one measurable lesion
10. Adequate organ functions
11. Adequate venous access for APH
12. Non-hematological adverse events induced by previous treatment must have recovered to Grade ≤1 according to Common Terminology Criteria for Adverse Events (CTCAE), except for alopecia and peripheral neuropathy
13. Women of childbearing potential must agree to use an effective and reliable contraceptive method during 28 days prior to lymphodepletion to 1 year post infusion; Male patients who have not undergone vasectomy and have sexual activity with women of childbearing potential must agree to the use of a barrier contraceptive method since lymphodepletion to 1 year post infusion, and sperm donation is prohibited during the study
14. Women of childbearing potential must have negative serum human chorionic gonadotropin β (β-hCG) test result at screening and 48 hours prior to lymphodepletion

Exclusion Criteria:

1. Pregnant or lactating women
2. Human immunodeficiency virus (HIV) serology positive, or active hepatitis B virus (HBV)/hepatitis C virus (HCV)/Syphilis/Tuberculosis/ Coronavirus disease 2019 (COVID-19)
3. Central nerve system (CNS) metastasis must have received treatment and been neurologically stable for ≥2 months, not requiring anti-seizure medications and off steroids for ≥ 1 month prior to APH
4. Another primary malignancy within 3 years (with some exceptions for completely-resected early-stage tumors)
5. Subjects with extensive metastases, or more rapid tumor progression prior to lymphodepletion in comparison to screening, etc. which might not be appropriate for further study treatment judged by the investigators
6. Systematic autoimmune disorders requiring long-term systematic treatment
7. Previously treated with any genetically engineered modified T cell therapy or other cell and gene therapy (CGT)
8. History of organ transplant
9. Uncontrolled or active infection within 72 hours prior to screening, APH, LD, or within 5 days prior to infusion
10. Subjects with other serious diseases that may restrict them from participating in this study
11. Clinically significant CNS disorders, such as epilepsy, stroke, Parkinson disease, etc
12. Grade ≥ 2 hemorrhage within 30 days prior to screening, or in need of longterm anticoagulants
13. Active digestive ulcer or gastrointestinal (GI) bleeding within 3 months prior to screening
14. Not satisfying wash-out period for APH
15. Previously allergic or intolerable to JWTCR001 or its components
16. Unable or unwilling to comply with the study protocol, judged by the investigators
17. Other situations implying that the subject might not be appropriate to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of dose-limiting toxicities (DLTs) | 28 days
  Dose-limiting toxicity (DLT) is defined as an adverse event that occurred within 28 days after JWTCR001 infusion that met any of the following criteria. Any Grade ≥3 non-hematologic toxicity associated with JWTCR001 that has not resolved to Grade ≤2 within 7 days, excluding clinically insignificant abnormalities in laboratory indicators. Grade ≥3 hematological toxicities. Grade ≥3 anaphylaxis. Grade ≥3 infection did not resolve to Grade ≤2 within 7 days after anti-infective treatment. Grade ≥3 autoimmune toxicity during treatment. Grade ≥3 cytokine release syndrome (CRS) during treatment that did not resolve to Grade ≤2 within 72 hours. Grade ≥3 TCR-T cell-associated encephalopathy syndrome/immune effector cell-associated neurotoxicity syndrome (CRES/ICANS) that did not resolve to Grade ≤2 within 72 hours. Grade 5 events of any nonmalignant cause.
Rate and severity of adverse events (AEs) and severe adverse events (SAEs) | 2 years
  An AE is defined as any unfavorable and unintended sign, symptom, or disease (new or worsening) temporally associated with the use of study therapy, regardless of whether or not a causal relationship with the study therapy can be determined.
Rate and severity of clinically-significant abnormalities in laboratory testings | 2 years
  Clinically-significant abnormalities in laboratory testings.

SECONDARY OUTCOMES:
Copy number of the vector transgene of JWTCR001 in peripheral blood | 2 years
  The pharmacokinetic parameters of JWTCR001 will be evaluated by quantitative polymerase chain reaction (qPCR) for the copy number of the vector transgene of JWTCR001 in peripheral blood to evaluate T-cell expansion and persistence.
MAGE-A4 specific TCR+ T Cell concentration of JWTCR001 in peripheral blood | 2 years
  The pharmacokinetic parameters of JWTCR001 will be evaluated by flow cytometry for the MAGE-A4 specific TCR+ T Cell concentration of JWTCR001 in peripheral blood to evaluate T cell expansion and persistence.
Antitumor efficacy-Progression-free survival (PFS) | 2 years
  The period from the day when the subject receives the infusion of cells to the first recorded tumor progression (whether treated or not) or death of any cause, which occurs first.
Antitumor efficacy-Duration of response (DOR) | 2 years
  The number of cases in which response are achieved from the start of cell infusion/the total number of evaluable cases (%).
Antitumor efficacy-Time to response (TTR) | 2 years
  The time from the first infusion to the first objective tumor response (tumor shrinkage of ≥30%) observed for patients who achieved a CR or PR.
Antitumor efficacy-Overall survival (OS) | 2 years
  The period from the first infusion to any cause of death.
Antitumor efficacy-Objective response rate (ORR) | 2 years
  The number of cases in which tumor size is reduced to complete response (CR) or partial response (PR) / the total number of evaluable cases (%). In the event of CR or PR, the subjects should confirm it no less than 4 weeks after the first evaluation.
Antitumor efficacy-Disease control rate (DCR) | 2 years
  The number of cases in which response are achieved from the start of cell infusion/the total number of evaluable cases (%).

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Department of GI Oncology,Peking University Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes